CLINICAL TRIAL: NCT05551403
Title: Electrophysiological Markers of Cortical Excitability to Predict Response to Treatment with Anti-seizure Medication - the ECORTA Study
Brief Title: Cortical Excitability and Treatment Response in People with Epilepsy
Acronym: eCORTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stichting Epilepsie Instellingen Nederland (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: NL77887.058.21; P21.092 (Other: METC LDD)
Record Dates: First submitted 2022-06-22; First posted 2022-09-22 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy
Keywords: Epilepsy; Transcranial Magnetic Stimulation; Evoked Potentials, Visual; Electroencephalography; Anticonvulsants; Seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rest-EEG, TMS-EEG/TMS-electromyography(EMG) and photic stimulation (Experimental)
  Interventions: Device: Eyes-closed rest-EEG registration; Device: Transcranial Magnetic Stimulation during EEG and EMG registrations; Device: Photic stimulation during eyes-closes EEG registration

INTERVENTIONS:
Device: Eyes-closed rest-EEG registration — Recording of spontaneous brain activity while eyes are shut for the duration of 7 minutes using a tablet with instructions
Device: Transcranial Magnetic Stimulation during EEG and EMG registrations — Recording of TMS-evoked EEG and EMG responses according to various stimulation protocols
Device: Photic stimulation during eyes-closes EEG registration — Recording of visual evoked potentials in the EEG during flash stimulation by light-emitting diode (LED) goggles (while eyes are closed)

SUMMARY:
Epilepsy is a medical condition marked by the occurrence of unpredictable, recurrent seizures. One-third of people with epilepsy continue to experience seizures, despite having attempted multiple forms of anti-seizure medication (ASM). Currently, response to ASM is assessed on a trial-and-error basis as their efficacy can only be determined in hindsight. This causes delays in finding the proper treatment per individual. Responsiveness of the outer brain layer to external stimuli, termed cortical excitability (CE), may be used as additional means of treatment evaluation.

In this study, the investigators aim to measure CE before and after starting with ASM, so as to determine whether indicators of CE can be used to predict favorable response to the medication. Participants in this study are adult individuals with uncontrolled seizures that will start with the novel anti-seizure medicine cenobamate. The investigators hypothesize that, after starting with ASM, the CE will decrease in people with epilepsy who show a favorable response to the medication. Conversely, the investigators anticipate that the CE will not decrease in those that do not react to the mediation.

The investigators will address this hypothesis by evaluating both brain activity (electroencephalography, EEG) during rest and during different types of stimulation (magnetic, light flashes). Besides, the investigators will measure the subjective experiences of participants by using questionnaires on the quality of life and feelings of anxiety or depression. These measurements are performed at a baseline instance, just before starting with ASM, and at two instances after start with the ASM. Participants in the study will track the occurrence of seizures - using a diary - from 12 weeks before ASM start up till 12 months after ASM start. The investigators will compare seizure frequency with both changes in brain activity and subjective experiences by the participants.

ELIGIBILITY:
Inclusion Criteria:

* In agreement with their own neurologist to initiate adjuvant treatment with cenobamate
* Diagnosed with refractory focal epilepsy, which means two ASMs failed to cause seizure freedom.
* Age of 18 years or older
* Having kept a seizure diary for the past 12 weeks
* At least one seizure in the past 12 weeks.

Exclusion Criteria:

* Photosensitive epilepsy
* Any device or structure in the skull or in close proximity of the head area containing metal, including cochlear implants, implanted neurostimulators, cardiac pacemakers and intracardiac lines.
* Persistent skull opening following trauma or surgery
* Evidence (clinical or radiological) of major structural abnormality of the motor cortex or pyramidal tracts
* Any major psychiatric condition such as a psychotic disorder
* Pregnancy
* Learning disabilities preventing the comprehension of oral and/or written instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Influence of cenobamate initiation on the resting motor threshold (rMT) when comparing short-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Pre- to post-cenobamate initiation change in cortical excitability assessed using the rMT in responders vs. non-responders. Classification into the latter is determined by comparing the seizure frequency in the 3 months post-target dose interval to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).
Influence of cenobamate initiation on transcranial magnetic stimulation (TMS)-evoked EEG potentials (TEP) when comparing short-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Pre- to post-cenobamate initiation change in cortical excitability assessed using TEP amplitudes in responders vs. non-responders. Classification into the latter is determined by comparing the seizure frequency in the 3 months post-target dose interval to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).

SECONDARY OUTCOMES:
Influence of cenobamate initiation on phase clustering and the neural network excitability index (NNEI) between visual evoked potential (VEP) trials when comparing short-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Pre- to post-cenobamate initiation change in cortical excitability assessed using VEP parameters (i.e. phase clustering and directly-related NNEI) in responders vs. non-responders. Classification into the latter is determined by comparing the seizure frequency in the 3 months post-target dose to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).
Influence of cenobamate initiation on the mean functional connectivity (MFC) and phase-amplitude coupling (PAC) in resting-state (rs-)EEG data when comparing short-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Pre- to post-cenobamate initiation change in cortical excitability using rs-EEG parameters (i.e. MFC and PAC values in the 0-120 Hz EEG frequency range) in responders vs. non-responders. Classification into the latter is determined by comparing the seizure frequency in the 3 months post-target dose interval to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).
Influence of cenobamate initiation on transcranial magnetic stimulation (TMS)-EMG and EEG, intermittent photic stimulation (IPS)-EEG and resting state (rs-)EEG parameters when comparing long-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2).
  TMS-EMG/-EEG parameters, IPS-EEG parameters, and rs-EEG parameters at T0, T1 and T2, incorporated as factors in a single multivariate statistical model alongside a factor for cenobamate response; i.e. responder or non-responder. Classification into the latter is determined by comparing the seizure frequency in the 12 months post-cenobamate initiation to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).
Correlation between the pre- to post-cenobamate initiation change in the resting motor threshold (rMT) and change in the seizure frequency when comparing short-term responders and non-responders to cenobamate | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Classification of subjects into responders and non-responders to cenobamate is determined by comparing the seizure frequency in the 3 months post-target dose interval to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).
Influence of cenobamate initiation on transcranial magnetic stimulation-induced EEG oscillations (TIO) when comparing short-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Pre- to post-cenobamate initiation change in cortical excitability assessed using TIO in responders vs. non-responders. Classification into the latter is determined by comparing the seizure frequency in the 3 months post-target dose interval to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).
Influence of cenobamate initiation on phase clustering between TEP trials when comparing short-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Pre- to post-cenobamate initiation change in cortical excitability assessed using phase clustering between TEP trials in responders vs. non-responders. Classification into the latter is determined by comparing the seizure frequency in the 3 months post-target dose interval to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).
Influence of cenobamate initiation on the neural network excitability index (NNEI) between TEP trials when comparing short-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Pre- to post-cenobamate initiation change in cortical excitability assessed using the NNEI between TMS-evoked EEG potential trials in responders vs. non-responders. Classification into the latter is determined by comparing the seizure frequency in the 3 months post-target dose to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).
Influence of cenobamate initiation on the short-interval intracortical inhibition (SICI) when comparing short-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Pre- to post-cenobamate initiation change in cortical excitability assessed using SICI of motor evoked potential amplitudes in responders vs. non-responders. Classification into the latter is determined by comparing the seizure frequency in the 3 months post-target dose interval to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).
Influence of cenobamate initiation on the long-interval intracortical inhibition (LICI) when comparing short-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Pre- to post-cenobamate initiation change in cortical excitability assessed using LICI of motor evoked potential amplitudes in responders vs. non-responders. Classification into the latter is determined by comparing the seizure frequency in the 3 months post-target dose interval to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).
Influence of cenobamate initiation on the cortical silent period (CSP) when comparing short-term responders and non-responders | At cenobamate initiation (T0), 7-8 weeks after cenobamate initiation (T1), and optionally at the maximum dose reached after individual treatment durations up to 1 year after cenobamate initiation (T2)
  Pre- to post-cenobamate initiation change in cortical excitability assessed using the CSP after motor evoked potentials in responders vs. non-responders. Classification into the latter is determined by comparing the seizure frequency in the 3 months post-target dose interval to the seizure frequency in the 3 months baseline interval (responder determined by a significant seizure reduction according to Poisson distribution statistics).

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Stichting Epilepsie Instellingen Nederland (SEIN), Heemstede, North Holland
  - Erasmus Medical Center, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No